CLINICAL TRIAL: NCT05386212
Title: National Taipei University of Nursing and Health Science
Brief Title: The Impact of an Instructional Web-based Healthcare App for Relieving Back Pain From Spinal Compression Fractures
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Cheng-Hsin General Hospital (Other)
Responsible Party: Principal Investigator, Pei-Hung Liao, Assistant Professor, National Taipei University of Nursing and Health Sciences
Other Study IDs: 108A-16
Record Dates: First submitted 2022-05-10; First posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Back Pain Lower Back Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control: regular nursing care instructions
  Interventions: Device: web app healthcare instructions for relieving back pain
- Expirement: web app healthcare instructions for relieving back pain
  Interventions: Device: web app healthcare instructions for relieving back pain

INTERVENTIONS:
Device: web app healthcare instructions for relieving back pain — This study designed web-based dynamic pain relief instructions for women with spinal compression fractures.

SUMMARY:
With the expected rise of patients with osteoporosis-induced fractures, it has become increasingly urgent to design and use specialized health education materials aimed at easing pain and improving bodily functions

DETAILED DESCRIPTION:
This study designed web-based dynamic pain relief instructions for women with spinal compression fractures. We collected patients' pain rating data the day before, one month after, and three months after providing the instructions.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women

Exclusion Criteria:

* postmenopausal women

Ages: 45 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — postmenopausal women
Study Population: postmenopausal women
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-05-12 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of back pain, and qualitative of life between groups | 3 months
  Follow-up observations of the control and experimental groups one month after the f intervention, as well as a significant difference between the data collected prior to the intervention and two months after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Hung Liao, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (3):
- Taiwan (3):
  - National Taipei university of nursing and health science, Taipei, Peito
  - Cheng Hsin General Hospital, Taipei
  - National Taipei university of nursing and health science, Taipei

IPD SHARING:
Plan to Share IPD: No